CLINICAL TRIAL: NCT07060417
Title: The Effects of SGLT2 Inhibition on Vascular Health and Physical Function in Veterans With CKD
Brief Title: Vascular Effects of SGLT2i in Non-diabetic CKD
Acronym: EMPA-CKD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEPH-006-24F
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Non-diabetic Chronic Kidney Disease
Keywords: CKD; SGLT2 inhibitor; endothelial function
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, phase-II study in 52 Veterans with non-diabetic CKD without heavy albuminuria (<300 mg/g) and eGFR 20-59 mL/min/1.73m2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization to either the placebo or empagliflozin group will be performed using a secure web-based system and allocation of empagliflozin vs. placebo in 1:1 ratio. The allocation of the study group will remain blinded to both participants and all study staff and investigators until the completion of the study. Participants will receive encapsulated empagliflozin and matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): The placebo will be encapsulated to look identical to the study drug.
  Interventions: Drug: Placebo
- Empagliflozin (Other): Matching 10-mg empagliflozin dose will be used.
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin 10 mg, encapsulated to match the placebo, will be used.
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — Matching placebo will be used.
  Arms: Placebo

SUMMARY:
Empagliflozin, a sodium-glucose co-transporter 2 inhibitor (SGLT2i), is a novel diabetic medication that reduces the risk of progression of chronic kidney disease (CKD) and heart failure and improves exercise tolerance regardless of the diabetes status. One of the important ways that empagliflozin improves health may be through its benefits on blood vessels. The effects of empagliflozin on blood vessels and physical function have not been examined in patients with chronic kidney disease, and it is less clear if empagliflozin may be beneficial in patients with chronic kidney disease without heavy urinary protein leakage. The investigators will examine if empagliflozin can improve blood vessel function and exercise tolerance in Veterans with chronic kidney disease without heavy urinary protein leakage.

DETAILED DESCRIPTION:
Overall Strategy: The investigators propose a randomized, double-blind, placebo-controlled, phase-II study in 52 Veterans with non-diabetic CKD without heavy albuminuria (<300 mg/g) and eGFR 20-59 mL/min/1.73m2 to investigate if empagliflozin, a selective SGLT2i, can improve vascular function, functional capacity, and plasma biomarkers of inflammation, oxidative stress, and nitric oxide (NO). Veterans will be recruited from the Salt Lake City VA and randomized to 10 mg of empagliflozin or placebo at 1:1 ratio and treated for 16 weeks.

Overarching Hypothesis: SGLT2 inhibition improves endothelial function in both macro- and micro-vasculature, in part, by mitigating inflammation and oxidative stress and augmenting NO bioavailability in patients with CKD, even in the absence of heavy albuminuria. The improved vascular function contributes to increased functional capacity.

Specific Aim 1: Comprehensively evaluate the efficacy of empagliflozin to improve vascular health, as determined by conduit artery endothelium-dependent vasodilation (flow-mediated dilation, FMD), peripheral microvasculature reactivity (passive limb movement, PLM), and arterial stiffness (carotid-femoral pulse wave velocity, PWV), in non-diabetic Veterans with CKD and albuminuria <300 mg/g.

Specific Aim 2: Evaluate the efficacy of empagliflozin to improve functional capacity using (a) handgrip exercise and (b) mobility tests (Timed Up-and-Go test, gait speeds, and 6-minute walk).

Specific Aim 3 (Exploratory): Evaluate the efficacy of empagliflozin to (a) reduce plasma biomarkers of systemic inflammation (C-reactive protein, interleukin-6, tumor necrosis factor- ) and oxidative stress (free radical concentration assessed by electron paramagnetic resonance spectroscopy) and (b) increase plasma NO, as reflected by plasma nitrite and nitrosyl hemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years of age or older
* eGFR 20-59 mL/min
* albuminuria <300 mg/g

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* expected to start dialysis or receive kidney transplantation or die within 4 months
* prior therapy with SGLT2i within the previous year
* unable to participate in the physical function tests (hand grip, walk)
* infections requiring intravenous antibiotic treatment
* malignancy requiring systemic therapy
* extremity skin ulceration requiring active therapy
* history of Fournier's gangrene
* severe hypoglycemia requiring external assistance within the past one year
* known allergy to empagliflozin
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in endothelium-dependent vasodilation as measured by flow mediated dilation (FMD) | baseline, 8 weeks, 16 weeks
  Brachial artery FMD will be used to assess if empagliflozin can improve endothelial function of conduit arteries in the upper limb. Brachial artery FMD outcome will be quantified as the maximal change in brachial artery diameter during the two-minute period after cuff release, expressed as a percentage increase from the pre-occlusion value (%FMD).

SECONDARY OUTCOMES:
Change in leg blood flow area-under-the-curve (LBF AUC) by Passive Leg Movement (PLM) | baseline, 8 weeks, 16 weeks
  PLM measures the movement-induced increase of blood flow mediated mostly by nitric oxide in feed arteries and microvascular beds of the leg. The total hyperemic response to PLM, expressed as LBF AUC, will be used as the main PLM endpoint.
Changes in aortic stiffness as measured by carotid-femoral pulse wave velocity (PWV) | baseline, 8 weeks, 16 weeks
  Carotid-femoral PWV is the gold standard for non-invasive assessment of central arterial stiffness, and our study will follow the established guidelines.
Changes in functional capacity as measured by handgrip exercise | baseline, 8 weeks, 16 weeks
  Handgrip strength will be measured during the maximal voluntary contraction using a handgrip dynamometer. The highest value of three maximal contractions will be used.
Mobility | baseline, 8 weeks, and 16 weeks
  Timed Up-and-Go test will be used to assess sequential mobility tasks that incorporate walking and turning. The gait speed test over a 10-meter distance will be assessed during both comfortable and fast-gait speeds. The 6-minute walk test will measure the total distance covered during a 6-minute duration.

OTHER OUTCOMES:
Changes in plasma biomarkers of systemic inflammation | baseline, 8 weeks, 16 weeks
  Assays for plasma TNF-alpha, CRP, IL-6 will be performed using a quantitative multiplex bead assay.
biomarkers of oxidative stress | baseline, 8 weeks, 16 weeks
  Plasma free radicals will be measured via electron paramagnetic resonance (EPR) spectroscopy. Measures
nitric oxide bioavailability | baseline, 8 weeks, 16 weeks
  Measures of NO bioavailability will be assessed using both nitrosyl-hemoglobin (NO-Hb) and ozone-chemiluminescence (Sievers Nitric Oxide Analyzer) methods for NO2-.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Cho, MD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No